CLINICAL TRIAL: NCT06991218
Title: Analysis of the Interaction Between Preoperative Lifestyle and Clinical Characteristics of Cardiac Surgery Patients and Perioperative Complications
Acronym: AKI
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-587; 2023YFC2506900 (Other Grant/Funding Number: National Key Research and Development Program of China)
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-05-27 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Cardiac Surgery; Hemoglobin; Perioperative Complications
Keywords: acute kidney injury; cardiac surgery; hemoglobin trajectory; Perioperative complications
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: The subjects of this study were patients aged 18 and above who underwent elective cardiac surgery.
  Interventions: Procedure: cardiac surgery

INTERVENTIONS:
Procedure: cardiac surgery — Adult patients (age ≥18 years) who underwent cardiac surgery with cardiopulmonary bypass were included.

SUMMARY:
Each year, over four million patients die within 30 days after surgery, accounting for 7.7% of global deaths. Due to its unique nature, cardiac surgery carries a significantly higher risk of perioperative complications and long-term mortality compared to non-cardiac surgeries. Therefore, the identification, management, and prevention of perioperative complications in cardiac surgery have long been a clinical focus. Common manifestations of perioperative organ injury include neurological complications, acute kidney injury, respiratory failure, gastrointestinal dysfunction, and liver injury. This study aims to explore the association between preoperative lifestyle and postoperative complications in cardiac surgery, as well as their interaction with clinical characteristics, in order to facilitate the prediction and prevention of perioperative complications. This retrospective cohort study plans to include adult patients undergoing elective cardiac surgery as the object of study. Different preoperative lifestyle habits will be considered as exposure factors to investigate the relationships between these exposure factors and the occurrence of major organ complications after cardiac surgery.

DETAILED DESCRIPTION:
The risk of death and major complications in patients undergoing general anesthesia is less than 1%, thanks to the implementation of clinical practice guidelines and checklists, as well as advancements in training, medications, monitoring devices, and equipment. Consequently, the safety of anesthesia has steadily improved over the past century. However, a recent assessment in Europe and the United States indicates that the overall postoperative mortality rate remains higher than expected and is considered the third leading cause of death globally, following ischemic heart disease and cancer. This statistical result should be noted, as perioperative deaths are multifactorial and it is challenging to clearly distinguish between surgery-related deaths and those attributed to preoperative comorbidities. Each year, over four million patients die within 30 days after surgery, accounting for 7.7% of global deaths.

Due to its unique characteristics, cardiac surgery carries a significantly higher risk of perioperative complications and long-term mortality compared to non-cardiac surgeries. Therefore, the identification, management, and prevention of perioperative complications in cardiac surgery have long been a clinical focus. Integrating surgical and patient-related risk factors in a personalized manner before, during, and after surgery can improve patient outcomes, as exemplified by Enhanced Recovery After Surgery (ERAS) protocols. However, despite improvements in all preventive measures, acute organ injury remains a common complication and a significant risk factor for morbidity and mortality in cardiac surgery patients. Common manifestations of perioperative organ injury include neurological complications, acute kidney injury (AKI), respiratory failure, gastrointestinal dysfunction, and liver injury.

Although much beneficial work has been done regarding the prevention and identification of perioperative complications in cardiac surgery, there is currently limited research on the impact of patients' preoperative medical history, personal history, and comorbidities on the occurrence and prediction of perioperative complications in cardiac surgery. This study focuses on exploring the association between preoperative lifestyle and postoperative complications in cardiac surgery. Additionally, the study will examine the interaction between preoperative laboratory tests and examinations, intraoperative anesthetic medication and vital sign monitoring, and preoperative lifestyle factors.

ELIGIBILITY:
1. Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patients scheduled for elective cardiac surgery.
3. Patients who received medical care at hospital from January 2018 to November 2022.

2.Exclusion Criteria:

1. Pregnant women.
2. Patients whose preoperative examinations indicated they had already met the diagnostic criteria for acute kidney injury (AKI) or acute respiratory distress syndrome (ARDS).
3. Patients with severe preoperative abnormalities in liver or kidney function.
4. Patients with more than 10% missing data in their basic clinical information.
5. Patients with mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥18 years) who underwent cardiac surgery with cardiopulmonary bypass in a large-scale comprehensive hospital between January 1, 2019 and October 31, 2023, were included.
Sampling Method: Probability Sample
Enrollment: 1366 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of perioperative complications of important organs | Within 30 days after the operation.
  The occurrence of perioperative complications of important organs (including the nervous system, respiratory system, urinary system, etc.)

SECONDARY OUTCOMES:
Acute kidney injury (AKI) | Within 7 days postoperatively.
  AKI was the primary outcome in this study, defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria as serum creatinine increase of ≥0.3 mg/dL within 48 hours postoperatively, or ≥1.5 times baseline creatinine within 7 days after surgery. AKI onset was determined on the first day when diagnostic criteria were met. Furthermore, AKI severity was staged according to following criteria: stage Ⅰ, serum creatinine increase of 0.3-4.0 mg/dL within 48 hours or 1.5-1.9 times baseline creatinine within 7 days postoperatively; stage Ⅱ, 2.0-2.9 times baseline creatinine within 7 days postoperatively; stage Ⅲ, serum creatinine increase >4.0 mg/dL within 48 hours or ≥3 times baseline within 7 days postoperatively.
Acute respiratory distress syndrome | Within 30 days after the operation.
  According to the 2012 Berlin definition, ARDS is classified into mild (PaO2/FiO2≤300mmHg), moderate (PaO2/FiO2≤200mmHg), or severe ARDS (PaO2/FiO2≤200mmHg).
Perioperative stroke | Within 30 days after the operation.
  CT within 30 days after the operation indicated hemorrhagic or ischemic cerebral infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Xuan Liu, Doctor, Principal Investigator — Department of Anesthesiology, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The relevant data need to be kept confidential.

REFERENCES:
- [Background] Glance LG, Lustik SJ, Hannan EL, Osler TM, Mukamel DB, Qian F, Dick AW. The Surgical Mortality Probability Model: derivation and validation of a simple risk prediction rule for noncardiac surgery. Ann Surg. 2012 Apr;255(4):696-702. doi: 10.1097/SLA.0b013e31824b45af. PMID 22418007
- [Background] Oprea AD, Del Rio JM, Cooter M, Green CL, Karhausen JA, Nailer P, Guinn NR, Podgoreanu MV, Stafford-Smith M, Schroder JN, Fontes ML, Kertai MD. Pre- and postoperative anemia, acute kidney injury, and mortality after coronary artery bypass grafting surgery: a retrospective observational study. Can J Anaesth. 2018 Jan;65(1):46-59. doi: 10.1007/s12630-017-0991-0. Epub 2017 Nov 2. PMID 29098634
- [Background] Section 2: AKI Definition. Kidney Int Suppl (2011). 2012 Mar;2(1):19-36. doi: 10.1038/kisup.2011.32. No abstract available. PMID 25018918
- [Background] Cao L, Ru W, Hu C, Shen Y. Interaction of hemoglobin, transfusion, and acute kidney injury in patients undergoing cardiopulmonary bypass: a group-based trajectory analysis. Ren Fail. 2022 Dec;44(1):1368-1375. doi: 10.1080/0886022X.2022.2108840. PMID 35946481
- See also: Definition and classification of AKI. — https://pubmed.ncbi.nlm.nih.gov/25018918/